CLINICAL TRIAL: NCT03833180
Title: A Phase 1 Dose-Escalation and Cohort-Expansion Study of VLS-101 in Subjects With Hematological Malignancies (waveLINE-001)
Brief Title: A Study of Zilovertamab Vedotin (MK-2140) (VLS-101) in Participants With Hematologic Malignancies (MK-2140-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VelosBio Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2140-001; VLS-101-0001 (Other: VelosBio)
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Diffuse Large B-cell Lymphoma; Richter Transformation Lymphoma; Burkitt Lymphoma; Lymphoplasmacytoid Lymphoma; T-cell Non-Hodgkin Lymphoma; Acute Lymphoid Leukemia; Acute Myeloid Leukemia; Waldenstrom Macroglobulinemia
Keywords: Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Leukemia, Lymphoid; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, Lymphoplasmacytoid; Waldenström Macroglobulinemia; Lymphoma, T-cell; Leukemia, Lymphoid, Acute; Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Leukemia, Lymphoid; Leukemia

STUDY DESIGN:
Intervention Model Description: Cohorts of 3 to 6 subjects will be sequentially enrolled at progressively higher dose levels within each dose schedule of zilovertamab vedotin using a 3+3 dose-escalation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Zilovertamab vedotin Schedule 1: Q1/3W (Experimental): Participants will be administered escalating doses of zilovertamab vedotin at 0.50, 1.00, 1.50, 2.25, 2.50, 2.75, and 3.00 mg/kg IV on Day 1 of repeated 21-day cycles (Q1/3W).
  Interventions: Drug: Zilovertamab vedotin
- Zilovertamab vedotin Schedule 2: Q2/3W (Experimental): Participants will be administered escalating doses of zilovertamab vedotin at 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, and 2.25 mg/kg IV on Day 1 and 8 of repeated 21-day cycles (Q2/3W).
  Interventions: Drug: Zilovertamab vedotin
- Zilovertamab vedotin Schedule 3: Q3/4W (Experimental): Participants will be administered escalating doses of zilovertamab vedotin at 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, and 2.25 mg/kg IV on Day 1, 8, and 15 of repeated 21-day cycles (Q3/4W).
  Interventions: Drug: Zilovertamab vedotin

INTERVENTIONS:
Drug: Zilovertamab vedotin — Zilovertamab vedotin administered via IV infusion per Schedule 1, 2, or 3 according to participant allocation.
  Other Names: VLS-101; MK-2140

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, immunogenicity, and efficacy of zilovertamab vedotin given intravenously (IV) across a range of dose levels in participants with previously treated hematological cancers including acute lymphocytic leukemia (ALL), acute myeloid leukemia (AML), Burkitt lymphoma (BL), chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), Richter transformation lymphoma (RTL), and T-cell non-Hodgkin lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* Men or women of age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Histological diagnosis of CLL/SLL, MCL, FL, MZL, DLBCL, RTL, BL, LPL/WM, T-cell NHL, ALL, or AML as documented in medical records.
* Hematological cancer under study has been previously treated and has progressed during or relapsed after prior systemic therapy.
* Hematological cancer is unlikely to be responsive to established therapies known to provide clinical benefit or the study candidate has developed an intolerance to established therapies known to provide clinical benefit.
* Presence of measurable cancer including CLL/SLL, MCL, FL, MZL, DLBCL, RTL, BL, LPL/WM, T-cell NHL, ALL, and AML.
* Current medical need for therapy due to disease-related symptoms or complications, cytopenias, lymphadenopathy, organomegaly, extranodal organ involvement, or progressive disease.
* Availability of pretreatment tumor tissue.
* Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥1 week before the start of study therapy.
* All acute toxic effects of any prior antitumor therapy (not including hydroxyurea, cytarabine, and/or cyclophosphamide used in subjects with acute leukemia) resolved to ≤Grade 1 before the start of study therapy (with the exception of alopecia [Grade 1 or 2 permitted] or selected laboratory parameters [Grade 1 or Grade 2 permitted with exceptions.
* Adequate bone marrow function.
* Adequate hepatic profile.
* Adequate renal function.
* Adequate coagulation profile.
* Negative antiviral serology.
* For female participants of childbearing potential, a negative serum pregnancy test.
* For both male and female participants, willingness to use protocol-recommended method of contraception from the start of the screening period until ≥6 months after the final dose of study therapy.
* Willingness and ability of the participant to comply with study activities.
* Evidence of a personally signed informed consent document.
* Previous treatment with an MMAE-containing drug is allowed.

Exclusion Criteria:

* Presence of malignancy involving the central nervous system.
* Presence of another cancer with disease manifestations or therapy that could adversely affect participant safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
* Significant cardiovascular disease within 3 months prior to start of study therapy.
* Significant screening electrocardiogram (ECG) abnormalities.
* Uncontrolled ongoing systemic bacterial, fungal, or viral infection.
* Known diagnosis of liver cirrhosis.
* Pregnancy or breastfeeding.
* Candidacy for hematopoietic stem cell transplantation (HSCT) or chimeric antigen receptor (CAR)-T-cell therapy with access to HSCT or CAR-T cells and a willingness to undergo such therapy.
* In participants with prior HSCT, evidence of graft-versus-host disease (GVHD) with Grade ≥2 serum bilirubin, Grade ≥3 skin involvement, or Grade ≥3 diarrhea.
* Prior solid organ transplantation.
* Major surgery within 4 weeks before the start of study therapy.
* Prior therapy with a receptor tyrosine kinase-like orphan receptor 1 (ROR1)-directed therapy.
* Has ongoing corticosteroid therapy (exceeding 30 mg daily of prednisone equivalent). Prednisone equivalent dosing must have been stable for at least 4 weeks prior to Cycle 1 Day 1 (C1D1). If corticosteroid treatment is required for lymphoma symptom control prior to C1D1, up to 100 mg per day of prednisone equivalent can be given for up to 5 days. In that case, all tumor assessments must have been completed prior to the start of corticosteroid treatment.
* Use of a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4.
* Use within 7 days prior to the start of study therapy of a drug known to prolong the QT interval.
* Concurrent participation in another therapeutic or imaging clinical trial.
* Presence of a medical condition that (in the judgement of the investigator) interferes with the ability of the participant to participate in the study.
* Has baseline peripheral neuropathy >Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of zilovertamab vedotin | Cycle 1 (Up to 21 Days)
  Participants will receive zilovertamab vedotin according to Schedule 1, 2, or 3. The MTD will be determined by the number of participants who experience a dose limiting toxicity (DLT). The MTD will be defined as the highest tested dose level at which ≥6 participants have been treated and which is associated with a Cycle 1 DLT in ≤17% of the participants.
Recommended Dosing Regimen (RDR) | Cycle 1 (Up to 21 Days)
  Selection of the RDR will be based on consideration of short- and long-term safety information together with available pharmacokinetic, pharmacodynamic, and efficacy data. The RDR may be the MTD or may be a lower dose within the tolerable dose range.

SECONDARY OUTCOMES:
Average number of zilovertamab vedotin infusions administered | Up to 5 months
  Zilovertamab vedotin drug administration will be assessed by prescribing records and the average number of zilovertamab vedotin infusions administered will be determined.
Number of participants with a treatment-emergent adverse event (TEAE) | Up to approximately 3.5 years
  An AE is any untoward medical occurrence in a participant administered a medicinal product; the event does not necessarily have a causal relationship with study drug administration or usage. Laboratory abnormalities, vital sign/oxygen saturation abnormalities, and adverse electrocardiogram (ECG) findings will also be recorded as AEs. A TEAE is defined as an AE that occurs or worsens in the period from the first dose of study drug administration to 30 days after the final dose of study drug administration. The number of participants with a TEAE will be reported for each arm.
Number of participants with a DLT | Cycle 1 (Up to 21 Days)
  A DLT is defined as a protocol pre-specified TEAE that occurs in Cycle 1 of zilovertamab vedotin therapy and is considered drug-related. Failure to recover to baseline by ≥21 days from the last dose of study drug in the current cycle due to a drug-related TEAE is also considered a DLT. The number of participants with a DLT will be reported for each arm.
Number of participants with a serious adverse event (SAE) | Up to approximately 3.5 years
  An SAE is defined as an untoward medical occurrence that results in any of the following outcomes: death, life-threatening situation, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or other medically significant event.
Number of participants with an adverse event of special interest (AESI) | Up to approximately 3.5 years
  Prespecified AESIs for this study will include: Grade ≥3 infusion reactions, tumor lysis syndrome (TLS) of any grade, and Grade ≥3 peripheral neuropathy. The number of participants with an AESI will be reported for each arm.
Number of participants that discontinue study treatment due to an AE | Up to approximately 3.5 years
  An AE is any untoward medical occurrence in a participant administered a medicinal product; the event does not necessarily have a causal relationship with study drug administration or usage. The number of participants that discontinue study treatment due to an AE will be reported for each arm.
Number of participants that use supportive care or concomitant medications | Up to approximately 3.5 years
  The number of participants that use supportive care or concomitant medications will be reported for each arm.
Plasma concentration of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Plasma concentration of zilovertamab vedotin will be reported for each arm.
Plasma concentration of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Plasma concentration of total UC-961 antibody will be reported for each arm.
Plasma concentration of monomethyl auristatin E (MMAE) | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Plasma concentration of MMAE will be reported for each arm.
Maximum plasma concentration (Cmax) of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Cmax of zilovertamab vedotin.
Time to maximum plasma concentration (Tmax) of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Tmax of zilovertamab vedotin.
Area under the plasma concentration time curve (AUC) of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine AUC of zilovertamab vedotin.
Volume of distribution (Vd) of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Vd of zilovertamab vedotin.
Clearance (CL) of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine CL of zilovertamab vedotin.
Apparent terminal half-life (t½) of plasma concentration of zilovertamab vedotin | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine t1/2 of plasma concentration of zilovertamab vedotin.
Cmax of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Cmax of total UC-961 antibody.
Tmax of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Tmax of total UC-961 antibody.
AUC of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine AUC of total UC-961 antibody.
Vd of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Vd of total UC-961 antibody.
CL of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine CL of total UC-961 antibody.
t1/2 of plasma concentration of total UC-961 antibody | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine t1/2 of plasma concentration of total UC-961 antibody.
Cmax of MMAE | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Cmax of MMAE.
Tmax of MMAE | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Tmax of MMAE.
AUC of MMAE | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine AUC of MMAE.
Vd of MMAE | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine Vd of MMAE.
CL of MMAE | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine CL of MMAE.
t1/2 of plasma concentration of MMAE | Cycle 1 Day 1, 2, 3, 8, 15: predose, end of infusion (up to 4 hours); Day 1, Day 8 (Schedule 2, 3), Day 15 (Schedule 3) of Cycles 2 through end of therapy (up to ~3.5 years): predose, end of infusion
  Blood samples collected predose and at multiple timepoints postdose will be used to determine t1/2 of plasma concentration of MMAE.
Number of participants with zilovertamab vedotin-reactive antibodies | Day 1 of Cycles 1 through end of therapy (up to approximately 3.5 years): predose and end of infusion (up to ~30 minutes)
  Number of participants with zilovertamab vedotin-reactive antibodies will be assessed.
Overall Response (OR) | Up to approximately 3.5 years
  OR will be defined by achievement of the following outcomes as indicated by disease type: CLL/SLL: Complete response (CR: disappearance of detectable disease per Cheson 2012 criteria), CR with incomplete blood count recovery (CRi: CR with ≥1 additional change in absolute neutrophil count, platelet count, or hemoglobin), partial response (PR: no evidence of new disease per Cheson 2012 criteria), or PR with lymphocytosis (PR except lack of decrease in peripheral blood absolute lymphocyte count); NHL: CR (disappearance of all detectable disease per Cheson 2014 criteria) or PR (≥50% decrease in the sum of the product of diameters of the index nodal and extranodal lesions); LPL/WM: CR, very good PR (CR with ≥90% decrease in M protein), PR, or minor response (criteria for PR or stable disease met per Cheson 2014); ALL: (CR, CRi, unconfirmed CR, or PR per National Comprehensive Cancer Network criteria); AML (CR, CRi, morphologic leukemia-free state [MLFS], or PR per Cheson 2003 criteria).
Complete Response without measurable residual disease (CRMRD-) | Up to approximately 3.5 years
  CRMRD- is defined as the achievement of ≤1 × 10^-4 malignant cells in bone marrow (as assessed by flow cytometry) in a participant who meets all other criteria for CR.
Percent change from baseline in tumor dimension | Up to approximately 3.5 years
  Percent change in tumor dimensions is defined as the percent change from baseline in the sum of the products of the diameters (SPD) of index lesions.
Time to Response (TTR) | Up to approximately 3.5 years
  TTR is defined as the interval from the start of study therapy to the first documentation of an objective response.
Duration of Response (DOR) | Up to approximately 3.5 years
  DOR is defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression/relapse or death from any cause.
Progression free survival (PFS) | Up to approximately 3.5 years
  PFS is defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression/relapse or death from any cause.
Time to Treatment Failure (TTF) | Up to approximately 3.5 years
  TTF failure is defined as the interval from start of study therapy to the earliest of the first documentation of disease progression/relapse, treatment failure (for participants with ALL or AML), the permanent cessation of study drug due to an AE, or death from any cause.
Overall Survival (OS) | Up to approximately 3.5 years
  OS is defined as the interval from the start of study therapy to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (14):
- United States (14):
  - City of Hope ( Site 0010), Duarte, California
  - University of California - San Diego ( Site 0003), La Jolla, California
  - UCLA Hematology & Oncology ( Site 0007), Los Angeles, California
  - University of Nebraska Medical Center ( Site 0006), Omaha, Nebraska
  - Northwell Health ( Site 0009), New Hyde Park, New York
  - Weill Cornell Medical College ( Site 0005), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0014), New York, New York
  - University of Rochester ( Site 0008), Rochester, New York
  - Memorial Sloan-Kettering Cancer Center ( Site 0019), Uniondale, New York
  - Oregon Health & Science University ( Site 0004), Portland, Oregon
  - MD Anderson Cancer Center ( Site 0001), Houston, Texas
  - MD Anderson Cancer Center ( Site 0011), Houston, Texas
  - University of Virginia Cancer Center ( Site 0012), Charlottesville, Virginia
  - Swedish Medical Center ( Site 0002), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wang ML, Barrientos JC, Furman RR, Mei M, Barr PM, Choi MY, de Vos S, Kallam A, Patel K, Kipps TJ, Rule S, Flanders K, Jessen KA, Ren H, Riebling PC, Graham P, King L, Thurston AW, Sun M, Schmidt EM, Lannutti BJ, Johnson DM, Miller LL, Spurgeon SE. Zilovertamab Vedotin Targeting of ROR1 as Therapy for Lymphoid Cancers. NEJM Evid. 2022 Jan;1(1):EVIDoa2100001. doi: 10.1056/EVIDoa2100001. Epub 2021 Oct 12. PMID 38319241
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/